CLINICAL TRIAL: NCT07162064
Title: Effectiveness and Safety of Heparinization for Radial Artery Occlusion After Transradial Cerebral Angiography in Patients With Acute Ischemic Stroke - A Multicenter, Prospective, Double-blind, Randomized Trail
Brief Title: Heparin for RAO Post-Transradial Angiography in AIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiang Luo (Other)
Responsible Party: Sponsor-Investigator, Xiang Luo, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-S021
Record Dates: First submitted 2025-08-26; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin Group (Experimental): Inject 2,500 units (2mL) of unfractionated heparin intra-arterially via sheath prior to angiography
  Interventions: Drug: Heparin - Therapeutic dosage
- Saline (0.9% NaCl) (Placebo Comparator): Inject 2ml saline intra-arterially via sheath prior to angiography
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Heparin - Therapeutic dosage — Intra-arterial sheath injection of heparin 2500 units before operation
  Arms: Heparin Group
Drug: Saline (0.9% NaCl) — Intra-arterial sheath injection of 2mL saline (0.9% sodium chloride)
  Arms: Saline (0.9% NaCl)

SUMMARY:
Cerebral angiography is a critical diagnostic tool in neurology, serving as the "gold standard" for evaluating cerebrovascular stenosis, hemodynamics, aneurysms, and arteriovenous malformations. Compared to the traditional transfemoral approach, transradial cerebral angiography (TRA) offers advantages such as preserved patient privacy, immediate post-procedure mobility, shorter hospitalization, and fewer access-site complications. Consequently, TRA has gained increasing acceptance among patients and clinicians as the preferred vascular access . However, radial artery occlusion (RAO) remains a common complication post-TRA, with reported incidence rates varying widely (1%-33%). RAO is particularly concerning as the radial artery serves as a key access for both cardiac and neurovascular interventions; its occlusion limits future procedural options.Evidence from interventional cardiology suggests that intra-arterial heparin administration significantly reduces RAO risk.However, patients undergoing transradial cerebral angiography are predominantly those with cerebrovascular diseases, including acute ischemic stroke (AIS)-a population at potential risk for hemorrhagic transformation.Although the 2022 Chinese Expert Consensus on Neurointerventional Diagnosis and Treatment via Transradial Access recommends intra-sheath heparin injection to prevent RAO, this recommendation is largely extrapolated from coronary intervention data. While several studies indicate that low-dose heparin is safe in moderate-to-severe AIS patients without increasing intracranial hemorrhage risk , high-level evidence specific to neurointerventional procedures-particularly in AIS patients-remains lacking.This multicenter, double-blind, randomized controlled trial (RCT) aims to: Evaluate the efficacy of intra-arterial heparin in preventing RAO following TRA cerebral angiography.Assess the safety of heparin in AIS patients, with a focus on hemorrhagic complications. By addressing these questions, the study will provide evidence-based guidance to optimize TRA outcomes, balancing RAO prevention with bleeding risk in neurovascular interventions. Its findings hold significant clinical value for improving the safety and efficacy of transradial cerebral angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Acute ischemic stroke onset within 7 days (inclusive)
3. Patients undergoing cerebral angiography via transradial approach
4. Participant or legal representative capable of providing informed consent

Exclusion Criteria:

1. Current anticoagulation therapy prior to procedure
2. Positive modified Allen's test result
3. History of coronary artery bypass grafting(CABG) with missing right radial artery graft
4. Severe forearm deformities (skin/musculoskeletal) or failed radial artery sheath placement
5. Suspected/confirmed pregnancy or lactation
6. Acute ischemic stroke with hemorrhagic transformation
7. Active systemic bleeding
8. Renal insufficiency (eGFR <30 mL/min or serum creatinine >200 μmol/L)
9. Investigator-determined ineligibility for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
24 hours radial artery occlusion rate after operation | 24 hours±12hours
  Radial artery occlusion rate was assessed by ultrasonography 24 hours±12hours after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SV, Cohen MG, Kandzari DE, Bertrand OF, Gilchrist IC. The transradial approach to percutaneous coronary intervention: historical perspective, current concepts, and future directions. J Am Coll Cardiol. 2010 May 18;55(20):2187-95. doi: 10.1016/j.jacc.2010.01.039. PMID 20466199
- [Background] Snelling BM, Sur S, Shah SS, Khandelwal P, Caplan J, Haniff R, Starke RM, Yavagal DR, Peterson EC. Transradial cerebral angiography: techniques and outcomes. J Neurointerv Surg. 2018 Sep;10(9):874-881. doi: 10.1136/neurintsurg-2017-013584. Epub 2018 Jan 8. PMID 29311120